CLINICAL TRIAL: NCT04791280
Title: Study of the Intestinal Microbiota of Patients With Systemic Sclerosis
Acronym: SCLEROMICROBIO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP201046
Record Dates: First submitted 2021-02-15; First posted 2021-03-10 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Systemic Sclerosis
Keywords: Gut microbiota; Systemic sclerosis
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with systemic sclerosis: On the day of inclusion, the faeces collection will be carried out by the patient using adapted equipment, either at the hospital or at home. In the case of a home collection, it will be carried out on the day of a planned hospital and preserved using equipment provided and tested to maintain the quality of the collection before storage.
  6 months after inclusion (+/- 2 months) a follow-up visit will be carried out and the patient will perform a second faecal sample.
  At the inclusion visit and at M6 the UCLA SCTC GIT 2.0 questionnaire will be completed by the patient.
  Interventions: Procedure: Faeces collection

INTERVENTIONS:
Procedure: Faeces collection — * faeces collection at inclusion
  * follow-up visit 6 months after inclusion

SUMMARY:
The term gut microbiota describes the entire intestinal microbial communities. Studies have established the important role played by the gut microbiome in modulating vital functions of the healthy host. The physiological effects of the microbiota for the host are, for the most part, beneficial. In several pathologies, an imbalance in the composition of the microbiota has been demonstrated.

Systemic sclerosis is an autoimmune, disorder of the connective tissue, characterized by vascular lesions, immunological abnormalities, and fibrosis of skin and internal organs As in many inflammatory diseases, there are painful digestive manifestations in systemic scleroderma that affect up to 90% of patients. The exact pathophysiology of the digestive involvement in systemic sclerosis is uncertain. The digestive manifestations of systemic sclerosis are frequent and can affect the entire digestive system.

However, there are few studies of the intestinal microbiota in this disease, which seems to be part of the same continuum of diseases with abnormalities of innate immunity. By analogy with chronic inflammatory bowel diseases, particularly Crohn's disease, we have raised the question of the existence of dysbiosis during scleroderma which could lead to episodes of acute, severe and recurrent inflammation of the peritoneum under the influence of triggering factors. The long-term prospects would be to look for ways to prevent attacks or to treat them more rapidly and effectively by using therapeutic targets in the intestinal microbiota.

The study population will be seen in the usual care setting, identically to all patients with systemic sclerosis treated in the department.

In case of an inflammatory disease outbreak, and depending on its severity, the patient will be seen again in consultation or hospitalized. Appropriate complementary examinations (biology, imaging, endoscopy) will be carried out and the treatment adapted.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Patient with a confirmed diagnosis of systemic sclerosis according to international criteria, before or after the start date of this study.
* Non-opposition of the patient

Exclusion Criteria:

* Subject under guardianship, curatorship or safeguard of justice
* Subject with state medical aid (AME)
* Subject does not speak French
* Subject unable to answer questions or express himself/herself
* Taking antibiotics or a colonic preparation within 6 weeks prior to stool collection will be a temporary contraindication to stool collection. The patient may be included, other usual care samples may be taken, but the stool sample will be deferred and taken at a later date.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with systemic sclerosis treated in the Internal Medicine Department of Saint Antoine Hospital and patients who will be newly diagnosed within 2 years after the beginning of the biological collection.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-03-31 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Prevalence of dysbiosis | Throughout the whole study, up to 6 months
  to study the prevalence of dysbiosis in patients with systemic sclerosis treated in the internal medicine department of St. Antoine Hospital in order to investigate prognostic biological parameters of disease progression, response to treatment and the occurrence of intestinal and extra-intestinal complications.

SECONDARY OUTCOMES:
Microbiota composition and diversity assessed by 16s sequencing | Throughout the whole study, up to 6 months
  To study the differences in microbiota according to the disease and its evolution under immunomodulating treatments.
The fecal bacterial composition in comparison to different subtypes of systemic sclerosis and evolution during the time | Throughout the whole study, up to 6 months
  To compare the markers of the intestinal microbiota between patients of this study and patients with IBD treated in in the Gastroenterology and Nutrition Department of St Antoine Hospital (existing biological collection SUIVITHEQUE).
Microbiota correlation | Throughout the whole study, up to 6 months
  To correlate microbiota abnormalities with disease progression, occurrence of intestinal and extraintestinal complications

CONTACTS AND LOCATIONS:
Overall Officials: Arsène MEKINIAN, professor, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Saint Antoine - service de médecine interne, Paris, France

IPD SHARING:
Plan to Share IPD: No